CLINICAL TRIAL: NCT07202143
Title: Methylprednisolone as Adjunct to Endovascular Thrombectomy for Acute Ischemic Stroke With Large Infarct Core and Post-stroke Lymphocytopenia -A Multicenter, Randomized, Double-blind, Placebo-controlled, Non-inferiority Trial
Brief Title: Methylprednisolone for Stroke With Large Infarct Core and Post-stroke Lymphocytopenia
Acronym: MIRACLE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: YiLin (Other)
Responsible Party: Sponsor-Investigator, YiLin, Deputy Director of Fujian Institute of Neurology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU [2025]887
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Large Infarct Core; Post-stroke Lymphocytopenia
MeSH Terms: interventions — Methylprednisolone Hemisuccinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone sodium succinate group (Experimental)
  Interventions: Drug: Methylprednisolone sodium succinate
- Methylprednisolone sodium succinate simulant (normal saline placebo) (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Methylprednisolone sodium succinate — Methylprednisolone sodium succinate Intravenous injection of methylprednisolone sodium succinate (Chongqing Lummy Pharmaceutical Co., Ltd., 40mg/ vial) with a dose of 2mg/kg (maximum dose of 160mg), once daily, for three consecutive days. The initial study drug will be administered as soon as possible after randomization. It is recommended that the initial study drug administrated before arterial access closure, but it should not be delayed more than 2 hours after arterial access closure.
  Arms: Methylprednisolone sodium succinate group
Drug: Normal Saline — Intravenous injection of placebo (normal saline) (Chongqing Lummy Pharmaceutical Co., Ltd., 40mg/ bottle) with a dose of 2mg/kg (maximum dose of 160mg), once daily, for three consecutive days. The initial study drug will be administered as soon as possible after randomization. It is recommended that the initial study drug administrated before arterial access closure, but it should not be delayed more than 2 hours after arterial access closure.
  Arms: Methylprednisolone sodium succinate simulant (normal saline placebo)

SUMMARY:
The efficacy and safety of early adjunctive methylprednisolone therapy in acute ischemic stroke patients with large infarct cores (ASPECTS score < 6) and post-stroke lymphocytopenia remain unclear. These immunocompromised patients face higher mortality rates and poorer clinical outcomes, with limited effective treatment options currently available. This multicenter, randomized, double-blind, placebo-controlled, non-inferiority trial aims to demonstrate that early methylprednisolone administration combined with reperfusion therapy is non-inferior to placebo in terms of survival and functional outcomes at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* The time from last known well to randomization was within 24 hours.
* Anterior circulation ischemic stroke was preliminarily determined according to clinical symptoms or imaging examination.
* Occlusion of the intracranial internal carotid artery, the M1- or M2-segment of the middle cerebral artery by confirmed by CT angiography (CTA), MR angiography (MRA), or digital subtraction angiography (DSA).
* Baseline National Institutes of Health Stroke Scale (NIHSS) ≥ 6.
* Baseline Alberta Stroke Program Early CT Score (ASPECTS) < 6 (based on non-contrast CT or MRI) or core infarct volume ≥ 50 ml (based on CTP with rCBF < 30%).
* Planned treatment with endovascular thrombectomy (EVT).
* Baseline peripheral blood lymphocyte < 0.8×10#/L
* Informed consent obtained from patients or their legal representatives.

Exclusion Criteria:

* Intracranial hemorrhage confirmed by cranial CT or MRI.
* mRS score > 2 before the time of last known well.
* Pregnant or lactating women.
* Allergic to contrast agents or glucocorticoids.
* Participating in other clinical trials.
* The artery is tortuous so that the thrombectomy device cannot reach the target vessel.
* Bleeding history (gastrointestinal and urinary tract bleeding) in recent 1 month.
* Chronic hemodialysis and severe renal insufficiency (glomerular filtration rate < 30 ml/min or serum creatinine > 220 umol/L [2.5 mg/ dL]).
* Life expectancy due to any advanced disease < 6 months.
* Follow-up is not expected to be completed.
* Intracranial aneurysm and arteriovenous malformation.
* Brain tumors with imaging mass effect.
* Systemic infectious disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 90 (±7) days | From randomization to 90 (±7) days
  Primary Efficacy Outcome. Defined as the number of any cause deaths observed divided by the number of subjects observed over the 90-day study period.

SECONDARY OUTCOMES:
Time from randomization to the occurrence of death from any cause at 90 (±7) days | From randomization to 90 (±7) days
  Secondary Efficacy Outcome; To evaluate death rate of the two treatment groups
mRS ordinal shift at 90 (±7) days (scores 5 and 6 are merged) | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 4 at 90 (±7) days | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 3 at 90 (±7) days | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 2 at 90 (±7) days | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Proportion of patients with mRS score 0 to 1 at 90 (±7) days or return to pre-stroke mRS score (for patients with prestroke mRS > 1) | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Midline shift at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome
Proportion of patients with midline shift maximum > 5 mm within 48 hours (%) | From randomization to 48 hours
  Secondary Efficacy Outcome
Relative hemispheric volume at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome
Net water uptake at 48 hours | From randomization to 48 hours
  Secondary Efficacy Outcome
Proportion of patients with decompressive craniectomy after EVT | From randomization until the date of discharge, an average of 1 week
  Secondary Efficacy Outcome
NIHSS score at 5-7 days or at early discharge | From randomization to 5-7 days (or at early discharge)
  Secondary Efficacy Outcome
EQ-5D-5L VAS at 90 (±7) days | From randomization to 90 (±7) days
  Secondary Efficacy Outcome
Proportion of patients with symptomatic intracranial haemorrhage (SICH) within 48 hours after EVT | From randomization to 48 hours
  Primary Safety Outcome. Based on the modified Heidelberg Bleeding Classification.
Proportion of patients with any intracranial haemorrhage (ICH) within 48 hours after EVT | From randomization to 48 hours
  Secondary Safety Outcome. Based on the modified Heidelberg Bleeding Classification.
Proportion of patients with pneumonia | From randomization until the date of discharge, an average of 1 week
  Secondary Safety Outcome
Proportion of patients with gastrointestinal haemorrhage within 7 days after EVT | From randomization to 7 days
  Secondary Safety Outcome
Incidence of any complications | From date of randomization until the date of discharge, an average of 1 week
  Secondary Safety Outcome
Incidence of any (serious) adverse events | From randomization to 90 (±7) days
  Secondary Safety Outcome

OTHER OUTCOMES:
mRS ordinal shift at 1 year (scores 5 and 6 are merged) | From randomization to 1 year
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 2 at 1 year | From randomization to 1 year
  Tertiary Efficacy Outcome
Proportion of patients with mRS score 0 to 1 at 1 year or return to pre-stroke mRS score (for patients with pre-stroke mRS > 1) | From randomization to 1 year
  Tertiary Efficacy Outcome
EQ-5D-5L VAS at 1 year | From randomization to 1 year
  Tertiary Efficacy Outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, the First Affiliated Hospital Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided